CLINICAL TRIAL: NCT04450797
Title: Intraoperative Ultrasound Guided Compared to Stereotactic Navigated Ventriculoperitoneal Shunt Placement: A Randomized Controlled Study
Brief Title: Intraoperative Ultrasound Guided Compared to Stereotactic Navigated Ventriculoperitoneal Shunt Placement
Acronym: NaVPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2019-02157; ch20Leu
Record Dates: First submitted 2020-06-22; First posted 2020-06-30 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Ventriculoperitoneal Shunt (VPS); Hydrocephalus
Keywords: Ventriculoperitoneal shunt (VPS)-dependency; VPS placement; Stereotactic Navigated Ventriculoperitoneal Shunt Placement; Ultrasound Guided (US-G) Ventriculoperitoneal Shunt Placement
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The primary outcome is the surgical intervention time, recorded by blinded anaesthesiologists. Some of the secondary outcomes (catheter placement (optimal vs. not optimal, grade I to IV), volumetry of side ventricles, Evans' Index) are measured by a blinded neuroradiologist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- US -G VPS placement (Active Comparator)
  Interventions: Device: US -G VPS placement, done by BK Medical 5000 US with burr hole probe (type 9063 N11C5S, 11-5 MHz).
- Stereotactic navigation for VPS placement (Active Comparator)
  Interventions: Device: Stereotactic navigation for VPS placement (Brainlab Dual Curve System with cranial navigation software version 3.1).

INTERVENTIONS:
Device: US -G VPS placement, done by BK Medical 5000 US with burr hole probe (type 9063 N11C5S, 11-5 MHz). — US -G VPS placement, done by BK Medical 5000 US with burr hole probe (type 9063 N11C5S, 11-5 MHz).
  Head not fixed, placed on horseshoe head holder, no preoperative navigation planning, catheter will be cut in length after positioning under real-time US guidance.
  Arms: US -G VPS placement
Device: Stereotactic navigation for VPS placement (Brainlab Dual Curve System with cranial navigation software version 3.1). — Stereotactic navigation for VPS placement (Brainlab Dual Curve System with cranial navigation software version 3.1).
  Head fixed in head clamp, entry point, trajectory and catheter length planned based on preoperative computer tomography imaging, catheter placed using navigated stylet.
  Arms: Stereotactic navigation for VPS placement

SUMMARY:
This study is to prospectively compare Ultrasound guided (US-G) Ventriculoperitoneal Shunt (VPS) placement to stereotactic navigation in a randomized controlled fashion with the surgical intervention time as primary outcome. All patients entering the University Hospital of Basel for elective or emergent VPS surgery will be randomized in 1:1 fashion to one of the study groups at admission or the day before the operation.

DETAILED DESCRIPTION:
Ventriculoperitoneal shunt (VPS) placement is one of the most frequent procedures in neurosurgical practice. The position of the proximal ventricular catheter is important since it influences possible malfunction of the VPS. For the improvement of accuracy in proximal VPS placement, navigation-based insertion techniques have been developed. VPS placement using stereotactic navigation has shown a high accuracy of catheter placement been developed. VPS placement using stereotactic navigation has shown a high accuracy of catheter placement, while the main limitations are that for referencing, the head of the patient needs to be fixed in a head holder and the preoperative set-up can be time-consuming. US-G VPS placement using a burr hole probe was described as an alternate for image-guided VPS placement technique. For US-G VPS placement head fixation or preoperative registration is not needed. This study is to prospectively compare Ultrasound guided (US-G) Ventriculoperitoneal Shunt (VPS) placement to stereotactic navigation in a randomized controlled fashion with the surgical intervention time as primary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Patients undergoing elective or emergent VPS placement (frontal or occipital shunt )

Exclusion Criteria:

* Revision surgery due to former VPS placement using the same side and location for VPS placement or when no complete shunt is revised (proximal and distal), resulting in a shorter operation time
* Ventriculoatrial or ventriculopleural Placement
* Women who are pregnant or breast feeding
* Intention to become pregnant during the course of the study
* Previous enrolment into the current study
* Enrolment of the investigator, his/her family members, employees, and other dependent persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2025-01-06 (Actual)

PRIMARY OUTCOMES:
surgical intervention time (minutes) | at Operation day (V2, up to 24 hours)
  time spent in the Operating Room (OR) by the surgeon, includes preparation time together (patient positioning, head clamping in the stereotactic navigation group) with the operation time of the neurosurgical part. Beginning ("positioning") and ending ("suture neurosurgical part") of this time interval is clearly defined and will be in a standardized manner recorded by blinded anaesthesiologists. . In the stereotactic navigation group, an additional 5 minutes will be added to the surgical intervention time for the preplanning of the navigation the day before the operation on the Brainlab workstation.

SECONDARY OUTCOMES:
Operation time (minutes) | at Operation day (V2, up to 24 hours)
  Operation time (minutes): time in minutes from "cut" to "suture"
Anaesthesia time (minutes) | at Operation day (V2, up to 24 hours)
  Anaesthesia time (minutes): time in minutes from "start anaesthesia" to "end anaesthesia"
Number of puncture attempts | at Operation day (V2, up to 24 hours)
  Number of puncture attempts
Catheter placement (optimal vs. not optimal) | at Operation day (V2,up to 24 hours), 2-3 days post-op. (V3), at discharge (V 4, approx. 7 days postop.), 6-8 weeks post-op (V5),6 months postop. (V6)
  Optimal catheter Placement: free-floating within the Cerebrospinal fluid (CSF) without touching ventricle wall or septum pellucidum, and the tip of the catheter located at the foramen of Monro showing an optimal length of the catheter. Catheters that did not fulfill all criteria have been defined as not optimal placed. Positioning of catheters will be further graded according to Yim et al. into grades I to IV (grade I: catheter terminates in the ipsilateral frontal horn, grade II: catheter terminates in contralateral frontal horn, grade III: catheter terminates in non-targeted CSF spaces, grade IV: catheter terminates intraparenchymally)
Change in volumetry of side ventricles | 1 day before Operation day (V1, up to 24 hours) and 2-3 days post-op. (V3)
  Change in volumetry of side ventricles pre- and postoperatively in cm3 (number and relative change)
Change in Evan's Index | before Operation day (V1) and 2-3 days post-op. (V3)
  Change in Evan's Index pre- and postoperatively (number and relative change).The Evans' index is the ratio of maximum width of the frontal horns of the lateral ventricles and the maximal internal diameter of the skull at the same level employed in axial CT images.
rate of complications (infection, bleeding, complications associated with navigation method) | from Operation day (V2, up to 24 hours) until 6 months postop. (V6)
  rate of complications (infection, bleeding, complications associated with navigation method)
mortality | from Operation day (V2, up to 24 hours) until 6 months postop. (V6)
  mortality
revision surgery (yes/no) | from Operation day (V2,up to 24 hours) until 6 months postop. (V6)
  revision surgery (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Severina Leu, Dr. med., Principal Investigator — Department of Neurosurgery, University Hospital of Basel; Luigi Mariani, Prof. Dr. med., Study Director — Department of Neurosurgery, University Hospital of Basel
Locations (1):
- Department of Neurosurgery, University Hospital of Basel, Basel, Switzerland

REFERENCES:
- [Derived] Leu S, Halbeisen F, Mariani L, Soleman J. Intraoperative ultrasound-guided compared to stereotactic navigated ventriculoperitoneal shunt placement: study protocol for a randomised controlled study. Trials. 2021 May 19;22(1):350. doi: 10.1186/s13063-021-05306-5. PMID 34011396